CLINICAL TRIAL: NCT02012387
Title: Multicenter Randomized, Double-blind, Placebo-controlled Parallel Clinical Trial to Assess Efficacy and Safety of Omalizumab (Xolair®) in a New Indication: Cholinergic Urticarial
Brief Title: Efficacy Study of Omalizumab in Cholinergic Urticaria
Acronym: CUN-OMAL-UCOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Hospital Universitari Joan XXIII de Tarragona. (Other); Hospital General Universitario Gregorio Marañon (Other); Complejo Hospitalario de Navarra (Other); Hospital Universitario Central de Asturias (Other); Hospital Clínico Universitario Lozano Blesa (Other); Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CUN-OMAL-UCOL
Record Dates: First submitted 2013-11-18; First posted 2013-12-16 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2017-04

CONDITIONS: Cholinergic Urticaria
Keywords: Cholinergic urticaria; Omalizumab
MeSH Terms: interventions — Exercise; Biological Products; Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active (Active Comparator): Omalizumab 300 mg Subcutaneous route 300 mg dose (independent from total IgE, weight or high)
  Interventions: Biological: Active
- Placebo (Placebo Comparator): Placebo Saline serum Subcutaneous route 0.6 ml saline serum with same volume as an active treatment
  Interventions: Biological: Placebo
- Open labeled (Active Comparator): After the double blinded period, all patients from both arms will receive the active drug for 8 more months.
  Interventions: Biological: Open labeled

INTERVENTIONS:
Biological: Active — Two injections will be administered every four weeks for four months, we will administer 4 doses within 16 weeks
  Other Names: Biological/Vaccine: Omalizumab; Other Names:; Xolair
  Arms: Active
Biological: Placebo — Two injections will be administered every four weeks for four months, we will administer 4 doses within 16 weeks
  Other Names: Biological/Vaccine: Placebo; Other Names: Saline serum
  Arms: Placebo
Biological: Open labeled — Two injections will be administered every four weeks for 8 months, we will administer 4 doses within 32 weeks
  Other Names: Biological: Omalizumab; Other Names:; Xolair
  Arms: Open labeled

SUMMARY:
To demonstrate the efficacy and safety of Omalizumab in a new indication, that is cholinergic urticaria.

DETAILED DESCRIPTION:
Physical urticarias, such as delayed pressure, cholinergic, dermatographism and cold urticaria, are highly disabling conditions[1]. Cholinergic urticaria occurs due to an active (e.g. exercise) or passive (e.g. hot bath) increase in core body temperature, causing itching and small hives with flare reaction on the trunk and limps that fade away upon cooling of the body[2].

As it is the case of chronic urticaria, physical urticarias have a great impact on patients' quality of life[3, 4]. However, these types of urticarias cause even more alteration on quality of life because of the limitations they cause in daily life activities, sports practicing[5] or work performance.

In spite of the high morbidity of this disease and the impact on quality of life, there is no available treatment. Antihistamines that usually control other types of urticaria could only partially alleviate cholinergic urticaria. There is only one paper[6] that shows efficacy doubling the dose of cetirizine above the recommended dosage on the Summary of Product Characteristics (off-label dosage). The poor response to antihistamine is justified by the minimal role of histamine in its physiopathology and only after employing very high doses[7].

The etiology and pathogenesis of hive formation remains unknown, though it is recognized that mast cells are clearly involved[8]. On the other hand, it seems that desensitization or tolerance could be induced in cholinergic urticaria[9]. Thus as it is the case of drug desensitization, Immunoglobulin E (IgE) receptor must also play a role in the development of this physical urticaria[10].

In the past years, the monoclonal humanized anti-IgE antibody (Omalizumab) was shown to be effective in control cholinergic urticaria[11] not respondent to conventional therapies at maximum or off-label doses. A negative response was also reported for cholinergic urticaria[12].

Our rationale for this approach in this type of urticaria is that Omalizumab exerts an inhibitory action on mast cell activation, as is the case of desensitization.

For that purpose, we will perform a multicenter, randomized, double-blind, placebo-controlled parallel clinical trial. We will include 24 patients including both female and male patients (age 14 years or older), non-respondent to antihistamines.

Efficacy will be evaluated through the negativization of the European Academy of Allergy and Clinical Immunology (EAACI), European Dermatology Forum (EDF) and urticaria network e.V (UNEV) standardized exercise challenge test, Visual Analog Scale (VAS), Chronic Urticaria Quality of Life validated questionnaire[13], patients' card of symptoms and use of rescue medication. Additional measures of efficacy will also be: the number of dropouts in each treatment group; the leave days due of urticaria and Emergency Department visits. Finally, safety will be assessed by means of recording and evaluation of adverse reactions during treatment.

As we previously stated, Omalizumab is not indicated for physical or other types of urticaria. The only indication is for treatment of moderate-to-severe allergic asthma. The hypothesis we are working on is that the monoclonal anti-IgE antibody Omalizumab could be as well effective in controlling physical urticaria symptoms in patients non-respondent to conventional therapy. We hypothesize that Omalizumab is able to revert the basophil or mast cell activation present in those urticaria types.

ELIGIBILITY:
Inclusion Criteria:

Adult female and male patients (age 14 years or older). Diagnosis of cholinergic urticaria trough clinical history and positive challenge test.

Non-respondent to supra therapeutic doses of antihistamines (defined as 2x the maximal dose included in the drug labeling) Written informed consent.

Exclusion Criteria:

Pruritus related to dermatitis or other skin condition. Any systemic disease that hampers follow up or interpretation of data. Omalizumab treatment within the previous 12 months. Any exclusion criteria included in the drug labeling. Any other conditions that do not allow the accomplishment of the clinical trial requisites, such as the abuse of drugs or alcohol.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Negativization of the exercise challenge test | It will be assessed prior to the study, and subsequently each 4 weeks up to 12 months.
  a. Our primary endpoint will be the negativization of the exercise challenge test: We will perform the exercise challenge test following the European Guidelines[14] for cholinergic urticaria. According with such guidelines, all centers will follow the same center standardized protocol. The patient will exercise in treadmill or running to the point of sweating and following for 15 more minutes, wearing warm clothing in a warm room. The test will be considered positive if exercise challenge leads to the typical rash over 10 minutes.

SECONDARY OUTCOMES:
Chonic Urticaria Quality of life | It will be evaluated up to 48 weeks.
  Quality of Life: QoL will be evaluated through the Spanish validated version of Chronic Urticaria quality of life (CU-Q2oL)
Patients' card | It will be assessed up to 48 weeks.
  Use of medication, VAS, daily symptoms, emergency visits, days off work.
Treatment drop offs in each sequence | Up to 48 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Departamento de Alergología. Clínica Universidad de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Background] Abajian M, Mlynek A, Maurer M. Physical urticaria. Curr Allergy Asthma Rep. 2012 Aug;12(4):281-7. doi: 10.1007/s11882-012-0269-0. PMID 22653630
- [Background] Hirschmann JV, Lawlor F, English JS, Louback JB, Winkelmann RK, Greaves MW. Cholinergic urticaria. A clinical and histologic study. Arch Dermatol. 1987 Apr;123(4):462-7. doi: 10.1001/archderm.123.4.462. PMID 3827277
- [Background] O'Donnell BF, Lawlor F, Simpson J, Morgan M, Greaves MW. The impact of chronic urticaria on the quality of life. Br J Dermatol. 1997 Feb;136(2):197-201. PMID 9068731
- [Background] Baiardini I, Giardini A, Pasquali M, Dignetti P, Guerra L, Specchia C, Braido F, Majani G, Canonica GW. Quality of life and patients' satisfaction in chronic urticaria and respiratory allergy. Allergy. 2003 Jul;58(7):621-3. doi: 10.1034/j.1398-9995.2003.00091.x. PMID 12823121
- [Background] Tlougan BE, Mancini AJ, Mandell JA, Cohen DE, Sanchez MR. Skin conditions in figure skaters, ice-hockey players and speed skaters: part II - cold-induced, infectious and inflammatory dermatoses. Sports Med. 2011 Nov 1;41(11):967-84. doi: 10.2165/11592190-000000000-00000. PMID 21985216
- [Background] Zuberbier T, Munzberger C, Haustein U, Trippas E, Burtin B, Mariz SD, Henz BM. Double-blind crossover study of high-dose cetirizine in cholinergic urticaria. Dermatology. 1996;193(4):324-7. doi: 10.1159/000246281. PMID 8993958
- [Background] Nakamizo S, Egawa G, Miyachi Y, Kabashima K. Cholinergic urticaria: pathogenesis-based categorization and its treatment options. J Eur Acad Dermatol Venereol. 2012 Jan;26(1):114-6. doi: 10.1111/j.1468-3083.2011.04017.x. Epub 2011 Mar 4. PMID 21371134
- [Background] Haas N, Toppe E, Henz BM. Microscopic morphology of different types of urticaria. Arch Dermatol. 1998 Jan;134(1):41-6. doi: 10.1001/archderm.134.1.41. PMID 9449908
- [Background] Kozaru T, Fukunaga A, Taguchi K, Ogura K, Nagano T, Oka M, Horikawa T, Nishigori C. Rapid desensitization with autologous sweat in cholinergic urticaria. Allergol Int. 2011 Sep;60(3):277-81. doi: 10.2332/allergolint.10-OA-0269. Epub 2011 Feb 25. PMID 21364312
- [Background] Morales AR, Shah N, Castells M. Antigen-IgE desensitization in signal transducer and activator of transcription 6-deficient mast cells by suboptimal doses of antigen. Ann Allergy Asthma Immunol. 2005 May;94(5):575-80. doi: 10.1016/S1081-1206(10)61136-2. PMID 15945561
- [Background] Metz M, Altrichter S, Ardelean E, Kessler B, Krause K, Magerl M, Siebenhaar F, Weller K, Zuberbier T, Maurer M. Anti-immunoglobulin E treatment of patients with recalcitrant physical urticaria. Int Arch Allergy Immunol. 2011;154(2):177-80. doi: 10.1159/000320233. Epub 2010 Aug 24. PMID 20733327
- [Background] Sabroe RA. Failure of omalizumab in cholinergic urticaria. Clin Exp Dermatol. 2010 Jun;35(4):e127-9. doi: 10.1111/j.1365-2230.2009.03748.x. Epub 2009 Nov 19. PMID 19925484
- [Background] Baiardini I, Pasquali M, Braido F, Fumagalli F, Guerra L, Compalati E, Braga M, Lombardi C, Fassio O, Canonica GW. A new tool to evaluate the impact of chronic urticaria on quality of life: chronic urticaria quality of life questionnaire (CU-QoL). Allergy. 2005 Aug;60(8):1073-8. doi: 10.1111/j.1398-9995.2005.00833.x. PMID 15969690
- [Background] Gaig P, Olona M, Munoz Lejarazu D, Caballero MT, Dominguez FJ, Echechipia S, Garcia Abujeta JL, Gonzalo MA, Lleonart R, Martinez Cocera C, Rodriguez A, Ferrer M. Epidemiology of urticaria in Spain. J Investig Allergol Clin Immunol. 2004;14(3):214-20. PMID 15552715